CLINICAL TRIAL: NCT03537872
Title: PROvide MIner-friendly SErvices for Integrated TB/HIV Care in Lesotho Study (PROMISE Study)
Brief Title: PROvide MIner-friendly SErvices for Integrated TB/HIV Care in Lesotho Study
Acronym: PROMISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Ministry of Health, Lesotho (Other Government); National University of Lesotho (NUL) (Unknown)
Responsible Party: Principal Investigator, Andrea Howard, Associate Professor of Epidemiology, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAR3789; U01GH002115 (NIH)
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: HIV
MeSH Terms: interventions — Public Sector

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Miner-Friendly (MF) Cohort (Experimental): Subjects will be enrolled over the 9-month enrollment period and will receive additional integrated strategies available at a miner-friendly service venue.
  Miner-Friendly (MF) Service Venues TB/HIV Integration Strategies.
  Interventions: Behavioral: Miner-Friendly (MF) Service Venues TB/HIV Integration Strategies
- Public Sector (PS) Cohort (Active Comparator): Subjects will be enrolled over the 9-month enrollment period and will receive the usual integrated care for the management of TB and HIV at a public sector health facility.
  Public Sector (PS) Health Facilities TB/HIV Integration Strategies
  Interventions: Behavioral: Public Sector (PS) Health Facilities TB/HIV Integration Strategies

INTERVENTIONS:
Behavioral: Miner-Friendly (MF) Service Venues TB/HIV Integration Strategies — In addition to the control condition strategies (marked "PS"), the MF intervention includes additional strategies (marked "MF"):
  STRUCTURAL LEVEL Co-location of TB and HIV services (PS); Co-location of clinical and non-clinical services (MF); Demand creation (MF); Weekend service hours (MF) CLINIC LEVEL Intensified TB case finding and IPT (PS); Test and START (PS); Training for healthcare workers (PS); Job aids and mentorship for healthcare workers (MF) INDIVIDUAL/FAMILY LEVEL Health literacy for patients (PS); Family counseling (PS - limited); One-way SMS text messaging and lay counselor support for adherence and retention (MF); A menu of options for medication refills for miners unable to visit the clinic on a monthly basis (MF)
  Other Names: MF intervention
  Arms: Miner-Friendly (MF) Cohort
Behavioral: Public Sector (PS) Health Facilities TB/HIV Integration Strategies — STRUCTURAL LEVEL Co-location of TB and HIV services CLINIC LEVEL Intensified TB case finding and IPT; Test and START; Training for healthcare workers INDIVIDUAL/FAMILY LEVEL Health literacy for patients; Family counseling (limited); Adherence support from nurses and village health workers
  Other Names: Control Condition (PS)
  Arms: Public Sector (PS) Cohort

SUMMARY:
The PROvide MIner-friendly SErvices for Integrated TB/HIV Care (PROMISE) study will assess the effectiveness, feasibility, and acceptability of integrated tuberculosis (TB)/HIV services provided in miner-friendly service venues in Lesotho that address barriers to early HIV diagnosis and antiretroviral therapy (ART) initiation, concurrent isoniazid preventive therapy (IPT), and retention in HIV care for migrant miners and their families in the context of President's Emergency Plan For AIDS Relief (PEPFAR) programming. The study will evaluate family-focused, integrated TB/HIV services for Basotho migrant miners and family members provided six days per week in miner-friendly service venues (MF), compared to public sector health facilities (PS), which will deliver usual integrated care for the management of TB and HIV.

The ultimate goals of the project are to 1) improve health outcomes among migrant miners and their families, a hard-to-reach population that represents a hotspot of TB/HIV transmission, in Lesotho and in PEPFAR programs more broadly; and 2) strengthen the implementation science research capacity of national and local institutions.

DETAILED DESCRIPTION:
TB is the most common opportunistic infection and a leading cause of death among people living with HIV (PLHIV). Early ART and IPT have been shown to reduce TB incidence, morbidity, and mortality among PLHIV, including those with high CD4 counts, and are recommended by the World Health Organization (WHO) as core strategies to reduce the burden of TB among PLHIV. Basotho migrant miners, who travel between their homes in Lesotho and work in South African mines, and their families are at elevated risk of HIV and TB, however, their testing, engagement, and retention in care and treatment are suboptimal. Implementation science research is urgently needed to determine an effective strategy for improving early detection of HIV and early initiation of ART and IPT among migrant miners and their families.

The PROMISE study is a mixed-methods implementation science study that will evaluate a miner-friendly intervention strategy to implement early ART and concurrent IPT for PLHIV. The study will assess the effectiveness, feasibility, and acceptability of integrated TB/HIV services for migrant miners and their family members provided in miner-friendly service venues (MF).

A prospective cohort study design will be used to evaluate the effectiveness of family-focused, integrated TB/HIV services for Basotho migrant miners and family members provided six days per week in miner-friendly service venues, compared to public sector health facilities (PS), which will deliver usual integrated care for the management of TB and HIV. All participants will be assessed at the time of HIV testing (baseline), and at months 3, 6, and 9.

Through implementing and measuring this enhanced TB/HIV service delivery model for miners and their families, study findings will have important implications on programs and policies broadly for PEPFAR, and specifically in Lesotho, for the organization and delivery of integrated TB/HIV services to migrant miners and their families. Findings will inform the development of more tailored interventions to promote HIV diagnosis, early ART, and IPT among miners with HIV, with possible implications for other types of mobile populations; enhance scientific awareness about the unique challenges facing miners in the context of their migration and high TB/HIV co-morbidity; and guide future efforts to develop differentiated service delivery models and integrated HIV/TB services in populations with a high prevalence of HIV and TB.

ELIGIBILITY:
MF Cohort Inclusion Criteria:

* Tested HIV-positive at MF site within one week of study enrollment
* Currently working or have worked in a South African mine, or are a family member of a miner (first-degree relative)
* Not on ART or IPT prior to testing HIV positive at the study site within the past week
* No history of IPT use
* 15 years or older
* Basotho origin
* Capacity for consent

MF Cohort Exclusion Criteria:

* Active TB
* Unwilling to provide a phone number or adhere to study procedures

PS Cohort Inclusion Criteria:

* Tested HIV-positive at either the OPD or voluntary counseling and testing (VCT) clinic on-site within one week of study enrollment
* Not on ART or IPT prior to testing HIV positive at the study site within the past week
* No history of IPT use
* 15 years or older
* Basotho origin
* Capacity for consent

PS Cohort Exclusion Criteria:

* Tested HIV-positive at other points of service, including antenatal clinic, labor & delivery, and TB clinics
* Active TB
* Unwilling to provide a phone number or adhere to study procedures

Health Care Provider Inclusion Criteria:

* 15 years or older
* Health care provider in MF or PS site
* Worked in the clinic for at least 3 months
* Capacity for consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of newly diagnosed HIV-positive participants initiated on ART (ART Initiation) | Up to 3 weeks after 9-month interview
  Participants will complete interviewer-administered questionnaires and data will be abstracted from their medical records to assess ART initiation. This is designed to determine if participants at MF are more likely to initiate ART compared to those at PS.
Proportion of newly diagnosed HIV-positive participants on ART initiated on IPT (IPT initiation) | Up to 3 weeks after 9-month interview
  Participants will complete interviewer-administered questionnaires and data will be abstracted from their medical records to assess IPT initiation. This is designed to compare if participants on ART at MF are more likely to initiate IPT compared to those at PS.

SECONDARY OUTCOMES:
CD4 count at enrollment | Up to 3 weeks after 9-month interview
  CD4 count at enrollment in care, collected from medical records.
Time to ART initiation | Up to 3 weeks after 9-month interview
  Time to ART initiation (in days) among newly diagnosed HIV-positive participants. Participants will complete interviewer-administered questionnaires and data will be abstracted from their medical records to assess ART initiation date.
Time to IPT initiation | Up to 3 weeks after 9-month interview
  Time to IPT initiation (in days) among newly diagnosed HIV-positive participants. Participants will complete interviewer-administered questionnaires and data will be abstracted from their medical records to assess IPT initiation date.
Proportion of newly diagnosed HIV-positive participants initiated on ART retained in care at 6 and 9 months at original clinic | Up to 3 weeks after 9-month interview
  ART retention, collected from medical records.
Proportion of newly diagnosed HIV-positive participants initiated on ART with plasma viral load <1000 copies/ml at 6 months after ART initiation | Up to 3 weeks after 9-month interview
  Viral suppression, collected from medical records.
Proportion of participants completed IPT among those who initiated IPT | Up to 3 weeks after 9-month interview
  IPT completion, collected from medical records.
Percentage of total prescribed doses of ART ingested, by self-report, averaged across study visits | Up to 9 months post baseline interview
  Participants will complete interviewer-administered questionnaires to assess ART adherence.
Percentage of positive IsoScreen tests at the first study visit after IPT initiation | Up to 9 months post baseline interview
  Participants will submit a urine sample which will be used to perform a IsoScreen test
Percentage of total prescribed doses of IPT ingested, by self-report, averaged across study visits | Up to 9 months post baseline interview
  Participants will complete interviewer-administered questionnaires to assess IPT adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea A. Howard, MD, MS, Principal Investigator — ICAP at Columbia University
Locations (5):
- Lesotho (5):
  - Maputsoe Filter Clinic, Hlotse
  - TEBA Leribe, Hlotse
  - TEBA Mafeteng, Mafeteng
  - Loretto Health Center, Maseru
  - TEBA Maseru, Maseru

IPD SHARING:
Plan to Share IPD: Yes
ICAP will make de-identified datasets from this project publically available, per CDC requirements.
  The dataset includes: 1) Routinely collected aggregate data from all patients undergoing HIV testing, including number tested for HIV, number testing HIV-positive, and number linked to care, stratified by sex and age; 2) Data collected from cohort participants in the miner-friendly service venue (MF) and public sector facility (PS) conditions, including a baseline interview, 3-, 6- and 9-month follow-up interviews, time-motion assessments, IsoScreen test results to measure adherence to IPT, and medical record abstraction of HIV clinic records; 3) Data collected from MF participants only, including in-depth interviews with miners and family members and health care providers; and 4) Data collected from all study sites, including a monthly site assessment of program characteristics and prospective data on service delivery costs.
Time Frame: Data will be available upon publication of the final report/major publication or 30 months after the completion of data collection, whichever comes first, per CDC requirements.
Access Criteria: Some data will be publically available.

REFERENCES:
- [Background] Lesotho Ministry of Health, ICF International. Lesotho Demographic and Health Survey 2014. Key Indicators Report. Maseru; 2015.
- [Background] Global tuberculosis report 2016. Geneva, Switzerland: World Health Organization; 2016.
- [Background] Howard AA, Saito S, Frederix K, Hirsch-Moverman Y, Maama LB, Tau P, et al. Integrating TB/HIV Services for Migrant Miners and Their Families in Lesotho. Conference on Retroviruses and Opportunistic Infections February 22-25, 2016. Boston. Abstract 738.
- [Background] Stuckler D, Basu S, McKee M, Lurie M. Mining and risk of tuberculosis in sub-Saharan Africa. Am J Public Health. 2011 Mar;101(3):524-30. doi: 10.2105/AJPH.2009.175646. Epub 2010 Jun 1. PMID 20516372
- [Background] Corbett EL, Marston B, Churchyard GJ, De Cock KM. Tuberculosis in sub-Saharan Africa: opportunities, challenges, and change in the era of antiretroviral treatment. Lancet. 2006 Mar 18;367(9514):926-37. doi: 10.1016/S0140-6736(06)68383-9. PMID 16546541
- [Background] Getahun H, Gunneberg C, Granich R, Nunn P. HIV infection-associated tuberculosis: the epidemiology and the response. Clin Infect Dis. 2010 May 15;50 Suppl 3:S201-7. doi: 10.1086/651492. PMID 20397949
- [Background] Charalambous S, Grant AD, Innes C, Hoffmann CJ, Dowdeswell R, Pienaar J, Fielding KL, Churchyard GJ. Association of isoniazid preventive therapy with lower early mortality in individuals on antiretroviral therapy in a workplace programme. AIDS. 2010 Nov;24 Suppl 5(0 5):S5-13. doi: 10.1097/01.aids.0000391010.02774.6f. PMID 21079429
- [Background] Durovni B, Saraceni V, Moulton LH, Pacheco AG, Cavalcante SC, King BS, Cohn S, Efron A, Chaisson RE, Golub JE. Effect of improved tuberculosis screening and isoniazid preventive therapy on incidence of tuberculosis and death in patients with HIV in clinics in Rio de Janeiro, Brazil: a stepped wedge, cluster-randomised trial. Lancet Infect Dis. 2013 Oct;13(10):852-8. doi: 10.1016/S1473-3099(13)70187-7. Epub 2013 Aug 16. PMID 23954450
- [Background] Golub JE, Pronyk P, Mohapi L, Thsabangu N, Moshabela M, Struthers H, Gray GE, McIntyre JA, Chaisson RE, Martinson NA. Isoniazid preventive therapy, HAART and tuberculosis risk in HIV-infected adults in South Africa: a prospective cohort. AIDS. 2009 Mar 13;23(5):631-6. doi: 10.1097/QAD.0b013e328327964f. PMID 19525621
- [Background] Golub JE, Saraceni V, Cavalcante SC, Pacheco AG, Moulton LH, King BS, Efron A, Moore RD, Chaisson RE, Durovni B. The impact of antiretroviral therapy and isoniazid preventive therapy on tuberculosis incidence in HIV-infected patients in Rio de Janeiro, Brazil. AIDS. 2007 Jul 11;21(11):1441-8. doi: 10.1097/QAD.0b013e328216f441. PMID 17589190
- [Background] Gupta A, Wood R, Kaplan R, Bekker LG, Lawn SD. Tuberculosis incidence rates during 8 years of follow-up of an antiretroviral treatment cohort in South Africa: comparison with rates in the community. PLoS One. 2012;7(3):e34156. doi: 10.1371/journal.pone.0034156. Epub 2012 Mar 30. PMID 22479548
- [Background] Samandari T, Agizew TB, Nyirenda S, Tedla Z, Sibanda T, Shang N, Mosimaneotsile B, Motsamai OI, Bozeman L, Davis MK, Talbot EA, Moeti TL, Moffat HJ, Kilmarx PH, Castro KG, Wells CD. 6-month versus 36-month isoniazid preventive treatment for tuberculosis in adults with HIV infection in Botswana: a randomised, double-blind, placebo-controlled trial. Lancet. 2011 May 7;377(9777):1588-98. doi: 10.1016/S0140-6736(11)60204-3. Epub 2011 Apr 12. PMID 21492926
- [Background] Yirdaw KD, Jerene D, Gashu Z, Edginton ME, Kumar AM, Letamo Y, Feleke B, Teklu AM, Zewdu S, Weiss B, Ruff A. Beneficial effect of isoniazid preventive therapy and antiretroviral therapy on the incidence of tuberculosis in people living with HIV in Ethiopia. PLoS One. 2014 Aug 8;9(8):e104557. doi: 10.1371/journal.pone.0104557. eCollection 2014. PMID 25105417
- [Background] INSIGHT START Study Group; Lundgren JD, Babiker AG, Gordin F, Emery S, Grund B, Sharma S, Avihingsanon A, Cooper DA, Fatkenheuer G, Llibre JM, Molina JM, Munderi P, Schechter M, Wood R, Klingman KL, Collins S, Lane HC, Phillips AN, Neaton JD. Initiation of Antiretroviral Therapy in Early Asymptomatic HIV Infection. N Engl J Med. 2015 Aug 27;373(9):795-807. doi: 10.1056/NEJMoa1506816. Epub 2015 Jul 20. PMID 26192873
- [Background] TEMPRANO ANRS 12136 Study Group; Danel C, Moh R, Gabillard D, Badje A, Le Carrou J, Ouassa T, Ouattara E, Anzian A, Ntakpe JB, Minga A, Kouame GM, Bouhoussou F, Emieme A, Kouame A, Inwoley A, Toni TD, Ahiboh H, Kabran M, Rabe C, Sidibe B, Nzunetu G, Konan R, Gnokoro J, Gouesse P, Messou E, Dohoun L, Kamagate S, Yao A, Amon S, Kouame AB, Koua A, Kouame E, Ndri Y, Ba-Gomis O, Daligou M, Ackoundze S, Hawerlander D, Ani A, Dembele F, Kone F, Guehi C, Kanga C, Koule S, Seri J, Oyebi M, Mbakop N, Makaila O, Babatunde C, Babatounde N, Bleoue G, Tchoutedjem M, Kouadio AC, Sena G, Yededji SY, Assi R, Bakayoko A, Mahassadi A, Attia A, Oussou A, Mobio M, Bamba D, Koman M, Horo A, Deschamps N, Chenal H, Sassan-Morokro M, Konate S, Aka K, Aoussi E, Journot V, Nchot C, Karcher S, Chaix ML, Rouzioux C, Sow PS, Perronne C, Girard PM, Menan H, Bissagnene E, Kadio A, Ettiegne-Traore V, Moh-Semde C, Kouame A, Massumbuko JM, Chene G, Dosso M, Domoua SK, N'Dri-Yoman T, Salamon R, Eholie SP, Anglaret X. A Trial of Early Antiretrovirals and Isoniazid Preventive Therapy in Africa. N Engl J Med. 2015 Aug 27;373(9):808-22. doi: 10.1056/NEJMoa1507198. Epub 2015 Jul 20. PMID 26193126
- [Background] World Health Organization. Guidelines for intensifed tuberculosis case-finding and isoniazid preventive therapy for people living with HIV in resource-constrained settings. Geneva; WHO 2010.
- [Background] WHO Policy on Collaborative TB/HIV Activities: Guidelines for National Programmes and Other Stakeholders. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK131887/ PMID 23586124
- [Background] World Health Organization. Policy brief: Consolidated guidelines on the use of antiretroviral drugs for treating and preventing HIV infection: What's new. November 2015. Geneva; WHO 2015.
- [Background] Lesotho Ministry of Health. Global AIDS response progress report 2015: Lesotho country report. Reporting period January-December 2014. Maseru; 2015.
- [Background] World Health Organization. Global tuberculosis control 2015. Geneva; WHO; 2015. http://www.who.int/tb/publications/global_report/gtbr15_main_text.pdf. Accessed Jan 20, 2016.
- [Background] Joint United Nations Programme on HIV/AIDS (UNAIDS). 90-90-90 An ambitious treatment target to help end the AIDS epidemic. http://www.unaids.org/sites/default/files/media_asset/90-90-90_en_0.pdf; Accessed March 22, 2016.
- [Background] PEPFAR Scientific Advisory Board (SAB). Recommendations Regarding Provision of ART for all Persons Living with HIV ("Test and START"). http://www.pepfar.gov/documents/organization/250048.pdf. Accessed March 21, 2016.
- [Background] Joint United States Programme on HIV/AIDS (UNAIDS). The GAP Report. Geneva; 2014. http://www.unaids.org/sites/default/files/media_asset/UNAIDS_Gap_report_en.pdf. Accessed Jul 18, 2015.
- [Background] Abdissa HG, Lemu YK, Nigussie DT. HIV preventive behavior and associated factors among mining workers in Sali traditional gold mining site Bench Maji zone, Southwest Ethiopia: a cross sectional study. BMC Public Health. 2014 Sep 26;14:1003. doi: 10.1186/1471-2458-14-1003. PMID 25256947
- [Background] Campbell C. Migrancy, masculine identities and AIDS: the psychosocial context of HIV transmission on the South African gold mines. Soc Sci Med. 1997 Jul;45(2):273-81. doi: 10.1016/s0277-9536(96)00343-7. PMID 9225414
- [Background] Corno L, de Walque D. Mines, migration and HIV/AIDS in southern Africa. J of African Economies 2012;21(3):465-498.
- [Background] International Organization for Migration. Country assessment on HIV prevention needs of migrants and mobile populations: Lesotho. Pretoria; 2010.
- [Background] Murray J, Davies T, Rees D. Occupational lung disease in the South African mining industry: research and policy implementation. J Public Health Policy. 2011;32 Suppl 1:S65-79. doi: 10.1057/jphp.2011.25. PMID 21730995
- [Background] Steele S. Human trafficking, labor brokering, and mining in southern Africa: responding to a decentralized and hidden public health disaster. Int J Health Serv. 2013;43(4):665-80. doi: 10.2190/HS.43.4.e. PMID 24397233
- [Background] Stuckler D, Steele S, Lurie M, Basu S. Introduction: 'dying for gold': the effects of mineral miningon HIV, tuberculosis, silicosis, and occupational diseases in southern Africa. Int J Health Serv. 2013;43(4):639-49. doi: 10.2190/HS.43.4.c. PMID 24397231
- [Background] Martins-Fonteyn E, Loquiha O, Wouters E, Raimundo I, Hens N, Aerts M, Meulemans H. HIV Susceptibility Among Migrant Miners in Chokwe: A Case Study. Int J Health Serv. 2016 Oct;46(4):712-33. doi: 10.1177/0020731415585988. Epub 2015 May 19. PMID 25995302
- [Background] Corbett EL, Watt CJ, Walker N, Maher D, Williams BG, Raviglione MC, Dye C. The growing burden of tuberculosis: global trends and interactions with the HIV epidemic. Arch Intern Med. 2003 May 12;163(9):1009-21. doi: 10.1001/archinte.163.9.1009. PMID 12742798
- [Background] Basu S, Stuckler D, Gonsalves G, Lurie M. The production of consumption: addressing the impact of mineral mining on tuberculosis in southern Africa. Global Health. 2009 Sep 29;5:11. doi: 10.1186/1744-8603-5-11. PMID 19785769
- [Background] Rees D, Murray J, Nelson G, Sonnenberg P. Oscillating migration and the epidemics of silicosis, tuberculosis, and HIV infection in South African gold miners. Am J Ind Med. 2010 Apr;53(4):398-404. doi: 10.1002/ajim.20716. PMID 19565628
- [Background] Corbett EL, Churchyard GJ, Clayton TC, Williams BG, Mulder D, Hayes RJ, De Cock KM. HIV infection and silicosis: the impact of two potent risk factors on the incidence of mycobacterial disease in South African miners. AIDS. 2000 Dec 1;14(17):2759-68. doi: 10.1097/00002030-200012010-00016. PMID 11125895
- [Background] Fielding KL, Grant AD, Hayes RJ, Chaisson RE, Corbett EL, Churchyard GJ. Thibela TB: design and methods of a cluster randomised trial of the effect of community-wide isoniazid preventive therapy on tuberculosis amongst gold miners in South Africa. Contemp Clin Trials. 2011 May;32(3):382-92. doi: 10.1016/j.cct.2010.12.008. Epub 2010 Dec 28. PMID 21193066
- [Background] Vynnycky E, Sumner T, Fielding KL, Lewis JJ, Cox AP, Hayes RJ, Corbett EL, Churchyard GJ, Grant AD, White RG. Tuberculosis control in South African gold mines: mathematical modeling of a trial of community-wide isoniazid preventive therapy. Am J Epidemiol. 2015 Apr 15;181(8):619-32. doi: 10.1093/aje/kwu320. Epub 2015 Mar 19. PMID 25792607
- [Background] Gilbert JA, Long EF, Brooks RP, Friedland GH, Moll AP, Townsend JP, Galvani AP, Shenoi SV. Integrating Community-Based Interventions to Reverse the Convergent TB/HIV Epidemics in Rural South Africa. PLoS One. 2015 May 4;10(5):e0126267. doi: 10.1371/journal.pone.0126267. eCollection 2015. PMID 25938501
- [Background] Kranzer K, van Schaik N, Karmue U, Middelkoop K, Sebastian E, Lawn SD, Wood R, Bekker LG. High prevalence of self-reported undiagnosed HIV despite high coverage of HIV testing: a cross-sectional population based sero-survey in South Africa. PLoS One. 2011;6(9):e25244. doi: 10.1371/journal.pone.0025244. Epub 2011 Sep 28. PMID 21969875
- [Background] Govender K, Akintola O, George G, Petersen I, Bhagwanjee A, Reardon C. Psychosocial and behavioural correlates of attitudes towards antiretroviral therapy (ART) in a sample of South African mineworkers. SAHARA J. 2011;8(2):55-64. doi: 10.1080/17290376.2011.9724986. PMID 23237682
- [Background] Bygrave H, Kranzer K, Hilderbrand K, Whittall J, Jouquet G, Goemaere E, Vlahakis N, Trivino L, Makakole L, Ford N. Trends in loss to follow-up among migrant workers on antiretroviral therapy in a community cohort in Lesotho. PLoS One. 2010 Oct 8;5(10):e13198. doi: 10.1371/journal.pone.0013198. PMID 20976289
- [Background] Barwise K, Lind A, Bennett R, Martins E. Intensifying action to address HIV and tuberculosis in Mozambique's cross-border mining sector. Int J Health Serv. 2013;43(4):699-719. doi: 10.2190/HS.43.4.g. PMID 24397235
- [Background] Currie CS, Williams BG, Cheng RC, Dye C. Tuberculosis epidemics driven by HIV: is prevention better than cure? AIDS. 2003 Nov 21;17(17):2501-8. doi: 10.1097/01.aids.0000096903.73209.ac. PMID 14600522
- [Background] Lesotho National TB Programme. Maseru; 2013.
- [Background] Baleta A. Southern African declaration targets TB in mining sector. Lancet. 2012 Oct 6;380(9849):1217-8. doi: 10.1016/s0140-6736(12)61698-5. No abstract available. PMID 23057075
- [Background] South African Development Community. Declaration on Tuberculosis in the Mining Sector. Maputo; 2012.
- [Background] Suphanchaimat R, Sommanustweechai A, Khitdee C, Thaichinda C, Kantamaturapoj K, Leelahavarong P, Jumriangrit P, Topothai T, Wisaijohn T, Putthasri W. HIV/AIDS health care challenges for cross-country migrants in low- and middle-income countries: a scoping review. HIV AIDS (Auckl). 2014 Feb 26;6:19-38. doi: 10.2147/HIV.S56277. eCollection 2014. PMID 24600250
- [Background] Lesotho Ministry of Health. A situation analysis of miners and ex-miners affected and infected by tuberculosis: Lesotho. Maseru; 2012.
- [Background] Dahab M, Charalambous S, Hamilton R, Fielding K, Kielmann K, Churchyard GJ, Grant AD. "That is why I stopped the ART": patients' & providers' perspectives on barriers to and enablers of HIV treatment adherence in a South African workplace programme. BMC Public Health. 2008 Feb 18;8:63. doi: 10.1186/1471-2458-8-63. PMID 18282286
- [Background] Siu GE, Wight D, Seeley J. How a masculine work ethic and economic circumstances affect uptake of HIV treatment: experiences of men from an artisanal gold mining community in rural eastern Uganda. J Int AIDS Soc. 2012 Jun 14;15 Suppl 1(Suppl 1):1-9. doi: 10.7448/IAS.15.3.17368. PMID 22713356
- [Background] Clinton Health Access Initiative. Health Findings and Recommendations: Domestic and Cross-Border Miners in Lesotho. Maseru; 2015.
- [Background] Nyamathi AM, Christiani A, Nahid P, Gregerson P, Leake B. A randomized controlled trial of two treatment programs for homeless adults with latent tuberculosis infection. Int J Tuberc Lung Dis. 2006 Jul;10(7):775-82. PMID 16848340
- [Background] Tavitian SM, Spalek VH, Bailey RP. A pharmacist-managed clinic for treatment of latent tuberculosis infection in health care workers. Am J Health Syst Pharm. 2003 Sep 15;60(18):1856-61. doi: 10.1093/ajhp/60.18.1856. PMID 14521037
- [Background] White MC, Tulsky JP, Goldenson J, Portillo CJ, Kawamura M, Menendez E. Randomized controlled trial of interventions to improve follow-up for latent tuberculosis infection after release from jail. Arch Intern Med. 2002 May 13;162(9):1044-50. doi: 10.1001/archinte.162.9.1044. PMID 11996616
- [Background] White MC, Tulsky JP, Menendez E, Arai S, Goldenson J, Kawamura LM. Improving tuberculosis therapy completion after jail: translation of research to practice. Health Educ Res. 2005 Apr;20(2):163-74. doi: 10.1093/her/cyg109. Epub 2004 Aug 16. PMID 15314035
- [Background] White MC, Tulsky JP, Menendez E, Goldenson J, Kawamura LM. Incidence of TB in inmates with latent TB infection: 5-year follow-up. Am J Prev Med. 2005 Nov;29(4):295-301. doi: 10.1016/j.amepre.2005.06.014. PMID 16242592
- [Background] Chaisson RE, Barnes GL, Hackman J, Watkinson L, Kimbrough L, Metha S, Cavalcante S, Moore RD. A randomized, controlled trial of interventions to improve adherence to isoniazid therapy to prevent tuberculosis in injection drug users. Am J Med. 2001 Jun 1;110(8):610-5. doi: 10.1016/s0002-9343(01)00695-7. PMID 11382368
- [Background] Tulsky JP, Pilote L, Hahn JA, Zolopa AJ, Burke M, Chesney M, Moss AR. Adherence to isoniazid prophylaxis in the homeless: a randomized controlled trial. Arch Intern Med. 2000 Mar 13;160(5):697-702. doi: 10.1001/archinte.160.5.697. PMID 10724056
- [Background] Durovni B, Cavalcante SC, Saraceni V, Vellozo V, Israel G, King BS, Cohn S, Efron A, Pacheco AG, Moulton LH, Chaisson RE, Golub JE. The implementation of isoniazid preventive therapy in HIV clinics: the experience from the TB/HIV in Rio (THRio) study. AIDS. 2010 Nov;24 Suppl 5(Suppl 5):S49-56. doi: 10.1097/01.aids.0000391022.95412.a6. PMID 21079428
- [Background] Diero L, Carter EJ, Silka A, Kimaiyo S, Gardner A, Yiannoutsos C, et al. The experience and outcomes of isoniazid preventive therapy in an HIV treatment program in Western Kenya. XVII International AIDS Conference 2008. Mexico City. Abstract MOAB0306; 2008.
- [Background] Sabapathy K, Van den Bergh R, Fidler S, Hayes R, Ford N. Uptake of home-based voluntary HIV testing in sub-Saharan Africa: a systematic review and meta-analysis. PLoS Med. 2012;9(12):e1001351. doi: 10.1371/journal.pmed.1001351. Epub 2012 Dec 4. PMID 23226107
- [Background] DiCarlo AL, Mantell JE, Remien RH, Zerbe A, Morris D, Pitt B, Abrams EJ, El-Sadr WM. 'Men usually say that HIV testing is for women': gender dynamics and perceptions of HIV testing in Lesotho. Cult Health Sex. 2014;16(8):867-82. doi: 10.1080/13691058.2014.913812. Epub 2014 May 22. PMID 24854495
- [Background] Shanaube K, Chaila JM, Floyd S, Schaap A, Griffith S, Hayes R, et al. Uptake of HIV Testing in the HPTN 071 (PopART) Trial in Zambia. Conference on Retroviruses and Opportunistic Infections February 22-25, 2016. Boston. Abstract 981.
- [Background] Barnighausen T, Chaiyachati K, Chimbindi N, Peoples A, Haberer J, Newell ML. Interventions to increase antiretroviral adherence in sub-Saharan Africa: a systematic review of evaluation studies. Lancet Infect Dis. 2011 Dec;11(12):942-51. doi: 10.1016/S1473-3099(11)70181-5. Epub 2011 Oct 24. PMID 22030332
- [Background] Lester RT, Ritvo P, Mills EJ, Kariri A, Karanja S, Chung MH, Jack W, Habyarimana J, Sadatsafavi M, Najafzadeh M, Marra CA, Estambale B, Ngugi E, Ball TB, Thabane L, Gelmon LJ, Kimani J, Ackers M, Plummer FA. Effects of a mobile phone short message service on antiretroviral treatment adherence in Kenya (WelTel Kenya1): a randomised trial. Lancet. 2010 Nov 27;376(9755):1838-45. doi: 10.1016/S0140-6736(10)61997-6. Epub 2010 Nov 9. PMID 21071074
- [Background] Pop-Eleches C, Thirumurthy H, Habyarimana JP, Zivin JG, Goldstein MP, de Walque D, MacKeen L, Haberer J, Kimaiyo S, Sidle J, Ngare D, Bangsberg DR. Mobile phone technologies improve adherence to antiretroviral treatment in a resource-limited setting: a randomized controlled trial of text message reminders. AIDS. 2011 Mar 27;25(6):825-34. doi: 10.1097/QAD.0b013e32834380c1. PMID 21252632
- [Background] Emenyonu N MW, Habyarimana J, Pops-Eleches C, Thirumurthy H, Ragland K, Bangsberg DR. Cash transfers to cover clinic transportation costs improve retention in care in a HIV treatment program in rural Uganda. 17th Conference on Retroviruses and Opportunistic Infections 16-19 February 2010. San Francisco. Abstract 831.
- [Background] El Sadr W, Branson B, Hall HI, Beauchamp G, Donnell D, Torian L, et al. Effect of financial incentives on linkage to care and viral suppression: HPTN 065 (TLC-Plus) Study. Conference on Retroviruses and Opportunistic Infections 23-26 February 2015. Seattle. Abstract 29.
- [Background] Etienne M, Burrows L, Osotimehin B, Macharia T, Hossain B, Redfield RR, Amoroso A. Situational analysis of varying models of adherence support and loss to follow up rates; findings from 27 treatment facilities in eight resource limited countries. Trop Med Int Health. 2010 Jun;15 Suppl 1:76-81. doi: 10.1111/j.1365-3156.2010.02513.x. PMID 20586964
- [Background] South African Development Community. Policy framework for population mobillity and communicable diseases in the SADC region. Gaborone; 2009.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] Group GGATSC. Tobacco Questions for Surveys: A Subset of Key Questions from the Global Adult Tobacco Survey (GATS), 2nd Edition. Atlanta, GA: Centers for Disease Control and Prevention; 2011.
- [Background] Kalichman SC, Simbayi LC, Jooste S, Toefy Y, Cain D, Cherry C, Kagee A. Development of a brief scale to measure AIDS-related stigma in South Africa. AIDS Behav. 2005 Jun;9(2):135-43. doi: 10.1007/s10461-005-3895-x. PMID 15933833
- [Background] Brock DM, Sarason IG, Sarason BR, Pierce GR. Simultaneous assessment of perceived global and relationship-specific support. Journal of Social and Personal Relationships 1996;13:143-152.
- [Background] Lubogo D, Ddamulira JB, Tweheyo R, Wamani H. Factors associated with access to HIV care services in eastern Uganda: the Kumi home based HIV counseling and testing program experience. BMC Fam Pract. 2015 Nov 3;16:162. doi: 10.1186/s12875-015-0379-6. PMID 26530286
- [Background] WHO Multi-Country Study on Women's Health and Domestic Violence: core questionnaire and WHO instrument, version 9. Geneva, Switzerland: World Health Organization; 2000.
- [Background] Dunkle KL, Jewkes RK, Brown HC, Yoshihama M, Gray GE, McIntyre JA, Harlow SD. Prevalence and patterns of gender-based violence and revictimization among women attending antenatal clinics in Soweto, South Africa. Am J Epidemiol. 2004 Aug 1;160(3):230-9. doi: 10.1093/aje/kwh194. PMID 15257996
- [Background] Wilson IB, Lee Y, Michaud J, Fowler FJ Jr, Rogers WH. Validation of a New Three-Item Self-Report Measure for Medication Adherence. AIDS Behav. 2016 Nov;20(11):2700-2708. doi: 10.1007/s10461-016-1406-x. PMID 27098408
- [Background] IsoScreen. Oxfordshire, UK: GFC Diagnostic Ltd.
- [Background] Whitfield R, Cope GF. Point-of-care test to monitor adherence to anti-tuberculous treatment. Ann Clin Biochem. 2004 Sep;41(Pt 5):411-3. doi: 10.1258/0004563041731637. PMID 15333195
- [Background] Guerra RL, Conde MB, Efron A, Loredo C, Bastos G, Chaisson RE, Golub JE. Point-of-care Arkansas method for measuring adherence to treatment with isoniazid. Respir Med. 2010 May;104(5):754-7. doi: 10.1016/j.rmed.2010.02.001. Epub 2010 Mar 3. PMID 20202806
- [Background] Mkopi A, Range N, Lwilla F, Egwaga S, Schulze A, Geubbels E, van Leth F. Adherence to tuberculosis therapy among patients receiving home-based directly observed treatment: evidence from the United Republic of Tanzania. PLoS One. 2012;7(12):e51828. doi: 10.1371/journal.pone.0051828. Epub 2012 Dec 19. PMID 23284782
- [Background] van den Boogaard J, Lyimo RA, Boeree MJ, Kibiki GS, Aarnoutse RE. Electronic monitoring of treatment adherence and validation of alternative adherence measures in tuberculosis patients: a pilot study. Bull World Health Organ. 2011 Sep 1;89(9):632-9. doi: 10.2471/BLT.11.086462. Epub 2011 May 20. PMID 21897483
- [Background] Patton MW. Developing a time motion study for a lean healthcare environment: University of Kentucky; 2011.
- [Background] Corbin J, Strauss A. Grounded theory research: Procedures, canons, and evaluative criteria. Qualitative Sociology 1990;13:3-21.
- [Background] Howard AA, Hirsch-Moverman Y, Frederix K, Daftary A, Saito S, Gross T, Wu Y, Maama LB. The START Study to evaluate the effectiveness of a combination intervention package to enhance antiretroviral therapy uptake and retention during TB treatment among TB/HIV patients in Lesotho: rationale and design of a mixed-methods, cluster-randomized trial. Glob Health Action. 2016 Jun 27;9:31543. doi: 10.3402/gha.v9.31543. eCollection 2016. PMID 27357074
- [Background] Howard AA, Hirsch-Moverman Y, Saito S, Gadisa T, Daftary A, Melaku Z. The ENRICH Study to evaluate the effectiveness of a combination intervention package to improve isoniazid preventive therapy initiation, adherence and completion among people living with HIV in Ethiopia: rationale and design of a mixed methods cluster randomized trial. Contemp Clin Trials Commun. 2017 Jun;6:46-54. doi: 10.1016/j.conctc.2017.03.001. Epub 2017 Mar 16. PMID 28626811
- [Background] Pathways to Engagement in HIV-Care for Newly Diagnosed South Africans, R01-MH83561, 2009-2014, Susie Hoffman DrPH, PI.

DOCUMENTS (1):
  • Informed Consent Form (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT03537872/ICF_000.pdf